CLINICAL TRIAL: NCT02707861
Title: A Phase 3, Multicenter, Expanded Access Study of Ibalizumab Plus an Optimized Background Regimen (OBR) in Treatment-Experienced Patients Infected With Multi-Drug Resistant (MDR) HIV-1
Brief Title: Ibalizumab Plus Optimized Background Regimen in Treatment-Experienced Patients With Multi-Drug Resistant HIV-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TaiMed Biologics Inc. (Industry)
Collaborators: Westat (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMB-311
Record Dates: First submitted 2016-03-08; First posted 2016-03-14 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: HIV
Keywords: HIV; Resistant; Salvage; ibalizumab; antibody; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — ibalizumab; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): IV ibalizumab (combined with optimized background regimen):
  800 mg once every two weeks for patients receiving that dosage on prior, successfully completed ibalizumab clinical trial
  OR
  2000 mg once every four weeks for patients receiving that dosage on prior, successfully completed ibalizumab clinical trial
  Administered for 48 weeks, or until ibalizumab becomes commercially available
  Interventions: Drug: ibalizumab; Drug: Optimized Background Regimen
- Cohort 2 (Experimental): IV ibalizumab (combined with optimized background regimen):
  800 mg once every two weeks for qualifying patients who have never received ibalizumab
  Administered for 48 weeks, or until ibalizumab becomes commercially available
  Interventions: Drug: ibalizumab; Drug: Optimized Background Regimen

INTERVENTIONS:
Drug: ibalizumab — Intravenous infusion of humanized monoclonal antibody binding with a region of Domain 2 of CD4 receptor, blocking post-attachment conformational changes necessary for HIV cell entry
  Other Names: TNX-355, Hu5A8
Drug: Optimized Background Regimen — An investigator-selected, standard-of-care combination regimen of antiretroviral agents for treating HIV-1 infection, selected based upon patient treatment history and the results of previous viral resistance testing. The combination must contain at least one agent other than ibalizumab to which the patient's virus is sensitive (susceptible).
  Other Names: antiretroviral therapy

SUMMARY:
Ibalizumab is a monoclonal antibody that works by blocking HIV entry into the immune system cells (CD4+ or T-cells) the virus typically infects. Ibalizumab is intended for use in combination with other anti-HIV drugs in people with multi-drug resistant HIV and limited treatment options. This study will collect further information on the safety and tolerability of intravenously administered (IV) ibalizumab combined with an optimized background regimen for treating multi-drug resistant HIV-1 infection, and will provide continuing access to ibalizumab for patients completing a prior ibalizumab clinical trial.

DETAILED DESCRIPTION:
Participants will enroll into one of two study cohorts. Cohort 1 will provide continued administration of IV ibalizumab for patients completing a prior ibalizumab clinical trial (TaiMed-sponsored or Investigator-Sponsored). Patients will continue to receive IV infusions of ibalizumab at the dosage assigned in the previous study - either 800 mg once every two weeks, or 2000 mg once every four weeks.

Cohort 2 will provide IV ibalizumab, 800 mg once every two weeks, for qualifying patients with multi-drug resistant HIV-1 and limited treatment options who have never previously received ibalizumab.

Participants may continue in this study for 48 weeks, or until ibalizumab becomes commercially available, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

(Cohort 1)

* Currently receiving ibalizumab via other TaiMed-sponsored or investigator-Sponsored protocol
* Are capable of understanding and have voluntarily signed the informed consent document

(Cohort 2)

* 18 years of age or older
* Are capable of understanding and have voluntarily signed the informed consent document
* Have documented HIV-1 infection by official, signed, written history (e.g., laboratory report), otherwise an HIV-antibody test will be performed
* Are able and willing to comply with all protocol requirements and procedures
* Have a viral load >1,000 copies/mL and documented resistance to at least one antiretroviral medication from each of three classes of antiretroviral medications as measured by previous viral resistance testing (resistance testing is not provided by the study for qualification purposes)
* Have a history of at least 6 months on antiretroviral treatment
* Are receiving a failing antiretroviral regimen OR have failed and are off therapy
* Have viral sensitivity/susceptibility to at least one antiretroviral agent, other than ibalizumab, as determined by previous resistance test performed within 6 months of screening and be willing and able to be treated with at least one agent to which the patient's viral isolate is fully sensitive/susceptible according to the resistance tests used for screening as a component of OBR
* If sexually active, are willing to use an effective method of contraception during the study and for 30 days after the last administration of the study drug

Exclusion Criteria:

(Cohort 1)

* There are no Exclusion Criteria for patients meeting the Inclusion Criteria for Cohort 1

(Cohort 2)

* Eligible for participation in other TaiMed-sponsored clinical trials of ibalizumab
* Any significant diseases (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, determined from screening, medical history and/or physical examination that, in the investigator's opinion, would preclude the patient from participating in this study
* Any significant acute illness within 1 week before the first administration of investigational medication on this study
* Any active infection secondary to HIV requiring acute therapy; however, patients that require maintenance therapy (i.e., secondary prophylaxis for opportunistic infections) will be eligible for the study.
* Any immunomodulating therapy (including interferon), systemic steroids, or systemic chemotherapy within 4 weeks before Day 0
* Any prior exposure to ibalizumab (formerly TNX-355 and Hu5A8)
* Any vaccination within 7 days before Day 0
* Any female patient who either is pregnant, intends to become pregnant, or is currently breastfeeding
* Any current alcohol or illicit drug use that, in the investigator's opinion, will interfere with the patient's ability to comply with the study schedule and protocol evaluations
* Any previous clinically significant allergy or hypersensitivity to any excipient in the ibalizumab formulation
* Any radiation therapy during the 28 days before first administration of investigational medication on this study
* Any clinically significant Grade 3 or 4 laboratory abnormality according to the Division of AIDS (DAIDS) grading scale, except for the following asymptomatic Grade 3 events:

  * triglyceride elevation
  * total cholesterol elevation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-03; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley T. Lewis, MD, MPH, Principal Investigator — TaiMed Biologics Inc.
Locations (32):
- United States (31):
  - Long Beach Education and Research Consultants, Long Beach, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Ruane Clinical Research Institute Inc., Los Angeles, California
  - Charles R. Drew University of Medicine and Science, Clinical and Translational Research Center, Los Angeles, California
  - Anthony Mills MD Inc., Los Angeles, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - eStudy Site, San Francisco, California
  - Kaiser Foundation Research Institute, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Fort Lauderdale, Florida
  - AIDS Healthcare Foundation - Kinder Medical Group, Miami, Florida
  - AIDS Healthcare Foundation - South Beach, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute, West Palm Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - University of Hawaii - John A. Burns School of Medicine, Honolulu, Hawaii
  - Howard Brown Health Center, Chicago, Illinois
  - National Institute of Allergy & Infectious Diseases, Bethesda, Maryland
  - ID Research Institute, Springfield, Massachusetts
  - Central West Clinical Research, St Louis, Missouri
  - AIDS Healthcare Foundation - Manhattan Midtown HCC, New York, New York
  - Chelsea Village Medical, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - East Carolina University, Greenville, North Carolina
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - St. Jude's Children's Research Hospital, Memphis, Tennessee
  - St. Hope Foundation Community Health Center, Bellaire, Texas
  - North Texas Infectious Disease Consultants, Dallas, Texas
  - Crofoot Research Center, Houston, Texas
  - Research Access Network, Houston, Texas
- Clinical Research PR, Inc., San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: IV ibalizumab (combined with optimized background regimen):
  800 mg once every two weeks for patients receiving that dosage on prior, successfully completed ibalizumab clinical trial
  OR
  2000 mg once every four weeks for patients receiving that dosage on prior, successfully completed ibalizumab clinical trial
  Administered for 48 weeks, or until ibalizumab becomes commercially available
  ibalizumab: Intravenous infusion of humanized monoclonal antibody binding with a region of Domain 2 of CD4 receptor, blocking post-attachment conformational changes necessary for HIV cell entry
  Optimized Background Regimen: An investigator-selected, standard-of-care combination regimen of antiretroviral agents for treating HIV-1 infection, selected based upon patient treatment history and the results of previous viral resistance testing. The combination must contain at least one agent other than ibalizumab to which the patient's virus is sensitive (susceptible).
- Cohort 2: IV ibalizumab (combined with optimized background regimen):
  800 mg once every two weeks for qualifying patients who have never received ibalizumab
  Administered for 48 weeks, or until ibalizumab becomes commercially available
  ibalizumab: Intravenous infusion of humanized monoclonal antibody binding with a region of Domain 2 of CD4 receptor, blocking post-attachment conformational changes necessary for HIV cell entry
  Optimized Background Regimen: An investigator-selected, standard-of-care combination regimen of antiretroviral agents for treating HIV-1 infection, selected based upon patient treatment history and the results of previous viral resistance testing. The combination must contain at least one agent other than ibalizumab to which the patient's virus is sensitive (susceptible).
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 41 | 38
Completed | 0 | 0
Not Completed | 41 | 38
Not completed — Went onto commercial drug | 30 | 23
Not completed — Adverse Event | 2 | 3
Not completed — Death | 5 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Physician Decision | 1 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (9.07) | 49.9 (11.7) | 51.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 37 | 34 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 16 | 28
  White | 27 | 20 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 2 | 4 | 6
  United States | 39 | 34 | 73
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 2 | 4 | 6
  United States | 39 | 34 | 73
Number of Study Participants Enrolled [Count of Participants; unit: Participants] | 41 | 38 | 79

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Ibalizumab + OBR
Description: Number of participants with Grade 3/4 adverse events possibly, probably, or definitely due to ibalizumab
Time Frame: Through 48 weeks
Population: intent-to-treat
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 41 | 38
participants | 8 | 9

2. Primary Outcome: Discontinuations Due to Adverse Events Related to Ibalizumab
Description: number of participants discontinuing ibalizumab treatment due to adverse events probably, possibly, or definitely related to ibalizumab
Time Frame: 48 weeks
Population: intent-to -treat
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 41 | 38
Participants | 0 | 3

3. Primary Outcome: Effectiveness of Ibalizumab + OBR (Cohort 2 Only)
Description: Number of patients in Cohort 2 achieving at least a 0.5 log change from Baseline in viral load at Day 7 of the study
Time Frame: 7 days
Population: As treated analysis
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 38
participants |  | 28

4. Secondary Outcome: Suppression to <50 Copies With Ibalizumab + OBR (Cohort 2 Only)
Description: Number of patients in Cohort 2 with HIV-1 RNA levels <50 copies/mL at week 48
Time Frame: 48 weeks
Population: as-treated-population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 17
Participants |  | 11

5. Secondary Outcome: Suppression to <400 Copies by Ibalizumab + OBR (Cohort 2 Only)
Description: Number of patients in Cohort 2 with HIV-1 RNA levels <400 copies/mL at week 48
Time Frame: 48 weeks
Population: as-treated-analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 17
Participants |  | 10

6. Secondary Outcome: Effectiveness of Ibalizumab + OBR by 1.0 Log10 Decrease in Viral Load From Baseline (Cohort 2 Only)
Description: Number of patients in Cohort 2 achieving at least a 1.0 log10 decrease in viral load from Baseline measurement at all assessment time points
Time Frame: 48 weeks
Population: as treated analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 17
Participants | 0 | 11

ADVERSE EVENTS:
Time Frame: Adverse event data is reported is reported for all subjects who received at least one dose of ibalizumab. The time period of observation ranges from day 1 to day 869 for study participants depending on the duration of ibalizumab therapy.
Description: The definitions of adverse events and methods of collection do not differ from clinical trials.gov definitions and methods.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 5/41 | 2/38
Serious Adverse Events (participants affected / at risk) | 16/41 | 15/38
Other Adverse Events (participants affected / at risk) | 39/41 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=41) | Cohort 2 (N=38)
sepsis (Infections and infestations) | 4 (4) | 4 (4)
cardiovascular disorder (Cardiac disorders) | 1 (1) | 1 (1)
DVT (Vascular disorders) | 3 (3) | 2 (2)
pneumonia (Infections and infestations) | 4 (4) | 4 (4)
acute renal failure (Renal and urinary disorders) | 2 (2) | 3 (3)
opportunistic infection (Infections and infestations) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=41) | Cohort 2 (N=38)
diarrhea (Gastrointestinal disorders) | 17 (17) | 10 (10)
headache (Nervous system disorders) | 8 (8) | 10 (10)
nausea (Gastrointestinal disorders) | 8 (8) | 9 (9)
rash (Skin and subcutaneous tissue disorders) | 17 (17) | 8 (8)

LIMITATIONS AND CAVEATS:
This trial included multiple populations- Cohort 1 included subjects who were treated with ibalizumab and OBR on previous trials including TMB-301, TMB-202, and 2 subjects on expanded access. The Cohort 2 subjects were subjects with MDR resistant virus who were treated with OBR plus ibalizumab. No subjects completed the planned duration of study as the vast majority were switched to commercial supply of drug when the drug was approved by USFDA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT02707861/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT02707861/SAP_001.pdf